CLINICAL TRIAL: NCT01096732
Title: Proof of Mechanism Study of an Oral Hedgehog Inhibitor (GDC-0449) in Patients With Resectable Pancreatic Ductal Adenocarcinoma in the Pre-operative Window Period
Brief Title: Hedgehog Inhibition for Pancreatic Ductal Adenocarcinoma (PDAC) in the Preoperative Setting (HIPPoS)
Acronym: HIPPoS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: Lisa Bax (Other)
Collaborators: Roche Pharma AG (Industry); Genentech, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Lisa Bax, Trial Coordinator, Cambridge University Hospitals NHS Foundation Trust
Organization: Cambridge University Hospitals NHS Foundation Trust (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OCRD 201014
Record Dates: First submitted 2010-03-30; First posted 2010-03-31 (Estimated); Last update posted 2014-01-08 (Estimated); Status verified 2014-01

CONDITIONS: Pancreatic Ductal Adenocarcinoma
Keywords: Pancreatic; adenocarcinoma; cancer
MeSH Terms: conditions — Adenocarcinoma; Neoplasms | interventions — HhAntag691

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GDC-0449 (Experimental): Study drug.
  Interventions: Drug: GDC-0449

INTERVENTIONS:
Drug: GDC-0449 — Gelatine capsules of 150mg.Taken O.D. for 14 days.
  Other Names: VISMODEGIB

SUMMARY:
This clinical trial is looking at the effect of a new drug called GDC-0449 in patients with cancer of the pancreas. Laboratory studies have shown that this drug blocks a process in pancreatic cells thought to be involved in cancer development and spread. This process is called the 'Hedgehog signalling pathway'. As yet, it is unclear whether blocking hedgehog signalling will directly affect the tumour cells themselves or the surrounding normal tissue. Understanding this distinction will help improve treatment strategies for pancreatic cancer. Patients will be offered to participate in this research study if they have localised pancreatic cancer that can be removed by surgery. In the period between diagnosis and surgery the investigators do not normally treat patients, however in this trial the investigators will ask patients to take GDC-0449 during the approximately two weeks until the day of surgery. All patients that enter this study will have undergone a diagnostic biopsy of the pancreatic tumour and the investigators will collect a second sample of the tumour at surgery. The main question of this study is whether the investigators can detect a change in hedgehog signalling in the normal tumour surrounding tissue. Furthermore the investigators will look very carefully whether this treatment is safe for patients. All problems before and after surgery will be carefully documented and the investigators have defined strict rules to stop the study if the investigators observe serious problems.

DETAILED DESCRIPTION:
Please contact Principal Investigators team for full details.

ELIGIBILITY:
Inclusion Criteria:

* Documented tissue diagnosis of pancreatic ductal adenocarcinoma with a sufficient amount of tissue for Laser Capture Micro-dissection (LCM) of the stromal and tumour compartments.
* Confirmed eligibility for a Whipple's or distal pancreatectomy procedure by Multi-Disciplinary Team (MDT) and surgeon review.
* Adequate organ function defined as:

  * Creatinine clearance ≥ 50ml/min (as defined by Cockcroft-Gault)
  * Electrolytes (Sodium (Na)/Potassium (K)/Calcium (Ca)) within institutional normal limits
  * Alanine transaminase (ALT)/Aspartate transaminase (AST) <5*ULN
  * Partial thromboplastin time (PTT)<2*ULN, prior supplementation with vitamin K is allowed
  * Adequate blood counts: neutrophils >1,500/μl, Hb > 6mmol/L,platelets >100.000/μl
  * Albumin ≥ 25mg/dL
* Written informed consent
* Male or female aged 18 years or over.
* World Health Organization (WHO) performance status 0-1
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.
* Males should not donate sperm during treatment or up to 3 months after the last dose.
* Women of childbearing potential are required to have a negative serum pregnancy test (with sensitivity of at least 25 mIU/mL) within 10-14 days and within 24 hours prior to the first dose of GDC-0449.

Exclusion Criteria:

* Known Hepatitis B/C or Human Immunodeficiency Virus (HIV) infection
* Known hypersensitivity to GDC-0449
* Active cardiac ischemic disease (this criterion only applies for participation in the imaging part of the study)
* Women, who are pregnant plan to become pregnant or are lactating (during the study or for up to 12 months after the last dose).
* Concurrent participation in another clinical trial using an investigational medicinal product.
* Other severe acute or chronic medical or psychiatric condition, or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or in the judgment of the investigator would make it undesirable for the patient to enter the trial (i.e. patients is not able to swallow tablets).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2011-02; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
To study the effect of GDC-0449 treatment on the stromal cell and tumour cell hedgehog signalling in patients with Pancreatic Ductal Adenocarcinoma. | 18 months
  1. To study the effect of GDC-0449 treatment on the stromal cell and tumour cell hedgehog signalling in patients with Pancreatic Ductal Adenocarcinoma.
  2. To study the safety and tolerability of pre-operative GDC-0449 treatment in patients who undergo Whipple's or distal pancreatectomy surgery for Pancreatic Ductal Adenocarcinoma.

CONTACTS AND LOCATIONS:
Overall Officials: David Tuveson, MD PhD, Principal Investigator — Cancer Research UK
Locations (1):
- Cambridge University Hospitals NHS Foundation Trust, Cambridge, United Kingdom